CLINICAL TRIAL: NCT02186535
Title: The Role of Vitamin D in Female Reproductive Tract Immunity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: A14-131
Record Dates: First submitted 2014-07-01; First posted 2014-07-10 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D; Calcium

ARMS (2):
- Daily dosing (Other): Daily oral capsule of Vitamin D in 4000 IU/day with daily oral capsules of 1000mg of calcium
  Interventions: Dietary Supplement: Vitamin D and Calcium
- weekly dosing (Other): Oral capsule Vitamin D 50,000 IU/week with a oral capsule of 1000mg of calcium, daily
  Interventions: Dietary Supplement: Vitamin D and Calcium

INTERVENTIONS:
Dietary Supplement: Vitamin D and Calcium

SUMMARY:
The purpose of this study is to assess the impact of approximately 8 weeks of Vitamin D (VitD) and calcium supplementation, using daily versus weekly supplementation regimens, on female reproductive tract immunity.

DETAILED DESCRIPTION:
This outpatient open label study will assess the impact of 8 weeks of daily versus weekly VitD and calcium supplementation on measures of cervicovaginal (CV) innate immune function, including antimicrobial and proinflammatory gene expression, Toll-like receptor (TLR)-mediated responses, immunohistochemical (IHC) analysis of immune cell markers, and microbiota in premenopausal women with insufficient serum VitD levels at baseline.

Women will be seen in 3 study visits and will be contacted by one scheduled follow-up telephone call after their final study visit. Volunteers will be consented at Visit 1 and undergo procedures to confirm they are eligible to continue in the study.

Once it has been confirmed that the participant meets all of the inclusion criteria and none of the exclusion criteria, baseline blood and genital samples will be taken in the luteal phase at Visit 2. The participant will then be given their first dose of VitD 4000 IU daily or 50,000 IU weekly in capsule form, which they will then administer for 8 weeks. Participants will also administer 1000 mg of calcium daily. Participants will return upon completion of supplementation for repeat of blood and genital samples (Visit 3).

ELIGIBILITY:
Inclusion Criteria:

* Serum 25(OH)D ≤ 25ng/mL (62 nmol/L)
* In good health, as evidenced by history and procedures at screening visits without any clinically significant systemic disease.
* Not at risk of an STI, meaning: In a monogamous heterosexual or same sex relationship with a partner who is not known to be HIV positive and has no known risks for STIs, or Sexually abstinent
* Willing and able to comply with study procedures
* 21 to 50 years of age
* Not at risk for pregnancy, meaning: Protected from pregnancy due to surgical sterilization of participant and or her sexual partner, Consistent condom use, In a same sex relationship or, Abstinent from sexual activity and planning to remain abstinent for the duration of the study
* Regular menstrual cycles (every 21 - 35 days) for the past two cycles, per participant report
* Willing to use sunscreen of SPF15 or higher when exposed to the sun for at least 15 minutes, and to avoid use of non-study Vitamin D, calcium, and multivitamin supplementation.

Exclusion Criteria:

* A clinically significant history of an abnormal Pap test (by written report) in the past year that has not been evaluated and/or treated, if indicated, according to standard guidelines
* Surgery or biopsy of the vagina or cervix within 14 days
* Current STI or lower genital tract infection including HIV-1, Chlamydia trachomatis (CT), Trichomonas vaginalis (TV), Neisseria Gonorrhoeae (NG), Hepatitis B, yeast vaginitis or bacterial vaginosis (BV) (by Nugent score of 7 - 10); this does not include asymptomatic HSV or human papilloma virus (HPV)
* Current presence of vulvar, anal and/or vaginal genital warts
* Current tobacco use of any amount
* Body Mass Index (BMI) of ≥ 35 kg/m2
* History of sensitivity/allergy to any component of the study product, topical anesthetic, or allergy to silver nitrate and/or Monsel's solution
* Known bleeding disorder that could lead to prolonged or continuous bleeding with biopsy, or taking anticoagulant drugs
* Grade 2 or higher laboratory abnormality, per the August 2009 update of the DAIDS Table for Grading the Severity of Adverse Events
* Systemic use in the last two weeks or anticipated use during the study of any of the following: corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs), antibiotics, anticoagulants or other drugs known to prolong bleeding and/or clotting, antifungals, antivirals (e.g., acyclovir or valacyclovir) or antiretrovirals (e.g., Viread). Note: Participants should avoid NSAIDS except for treatment of dysmenorrhea during menses. Participants may use acetaminophen on an as-needed but not daily basis during the study.
* Known risk factors for hypercalcemia (e.g. malignancy or granulomatous disease) or malabsorption syndromes (e.g. celiac disease, radiation enteritis, active inflammatory bowel disease).
* Other conditions that, in the opinion of the investigator, would constitute contraindications to participation in the study or would compromise the ability to comply with study protocols, such as any major chronic illness including but not limited to cancer, serious autoimmune disease, metabolic disorders or a major psychiatric disorder (e.g., schizophrenia)
* Current participation in any other drug or device study, or any study which, in the opinion of the investigator, would jeopardize interpretation of results of this study
* Use of depot medroxyprogesterone acetate (DMPA) in last six months
* Use of any other hormonal contraceptive method (oral, transdermal, transvaginal, implant, or intrauterine device) without 2 subsequent, normal menses since stopping hormonal contraceptives
* Current use of copper IUD
* Currently pregnant or pregnancy within the past 3 months
* Currently breastfeeding or having breastfed an infant in the last two months

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Vitamin D concentrations in serum and vaginal secretions | over 8 weeks of use
  Assess the impact of daily versus weekly Vitamin D and calcium supplementation regimens on Vitamin D concentrations in serum and on soluble markers innate mucosal immunity and inflammatory response in cervicovaginal secretions.

SECONDARY OUTCOMES:
Assessment of Gene Expression | over 8 weeks of use
  Assess gene expression of epithelial factors associated with innate immune response in CV tissues before and after VitD and calcium supplementation.
Assessment of immune cell activation and phenotype by IHC in CV tissues | over 8 weeks of use
  Assess immune cell activation and phenotype by IHC in CV tissues before and after VitD and calcium supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Thurman, M.D., Principal Investigator — CONRAD
Locations (1):
- Eastern Virginia Medical School CONRAD Clinical Research Center, Norfolk, Virginia, United States